CLINICAL TRIAL: NCT02162446
Title: An Open-label, Micro-dosing Study to Evaluate Safety, Biodistribution, Dosimetry and Preliminary Efficacy of Two Single 68Ga-OPS202 Doses for the Diagnostic Imaging of Somatostatin Receptor-positive Gastro-entero-pancreatic Neuroendocrine Tumors (GEP NET) Using Positron-emission Tomography / Computed Tomography (PET/CT)
Brief Title: 68Ga-OPS202 Study for Diagnostic Imaging of GEP NET
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPS-B-001; 2014-001881-88 (EudraCT Number)
Record Dates: First submitted 2014-06-03; First posted 2014-06-12 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 68Ga-OPS202 (Experimental): Satoreotide trizoxetan will be administered in two sequentially ascending peptide doses
  Interventions: Drug: satoreotide trizoxetan

INTERVENTIONS:
Drug: satoreotide trizoxetan
  Other Names: 68Ga-OPS202

SUMMARY:
The purpose of this study is to assess the safety and tolerability of 68Ga-OPS202 used for the diagnosis of gastroenteropancreatic neuroendocrine tumors (GEP NETs).

ELIGIBILITY:
Inclusion Criteria:

* A diagnostic CT or MRI of the tumor region within the previous 6 months prior to dosing day is available.
* A somatostatin receptor scan with results in the previous 6 months prior to dosing day.
* At least 1 lesion detected by the previous somatostatin receptor scan.
* Not exceeding 30 lesions / organ detected by the previous somatostatin receptor scan.
* Blood test results as follows (WBC: ≥ 3*109/L, Hemoglobin: ≥ 8.0 g/dL, Platelets: ≥ 50x109/L, ALT, AST, AP: ≤ 5 times ULN, Bilirubin: ≤ 3 times ULN)
* ECG: any abnormalities have to be clarified by a cardiologist.
* Serum creatinine: within normal limits or < 120 μmol/L for patients aged 60 years or older.
* Calculated GFR ≥ 45 mL/min.
* Negative pregnancy test in women capable of child-bearing.

Exclusion Criteria:

* Known hypersensitivity to 68Ga, to NODAGA, to JR11 or to any of the excipients of 68Ga-OPS202.
* History of, or current active allergic or autoimmune disease, including asthma or any condition requiring long-term use of corticosteroids.
* Presence of active infection at screening or history of serious infection within the previous 6 weeks.
* Known human immunodeficiency virus (HIV) or positive serology for HIV, hepatitis B and C.
* Any condition that precludes raised arms position for prolonged imaging purposes.
* Neuroendocrine tumor specific treatment between last somatostatin receptor imaging and start of this study. Exception is the therapeutic use of any somatostatin analog (see below).
* Therapeutic use of any somatostatin analog, including Sandostatin® LAR (within 28 days) and Sandostatin® (within 2 days) prior to study imaging. If a patient is on Sandostatin® LAR a wash-out phase of 28 days is required before the injection of the study drug. If a patient is on Sandostatin® a wash-out phase of 2 days is required before the injection of the study drug.
* Administration of another investigational medicinal product within 30 days prior to entry.
* Prior or planned administration of a radiopharmaceutical within 8 half-lives of the radionuclide used on such radiopharmaceutical including at any time during the current study.
* Current > grade 2 toxicity from previous standard or investigational therapies, per US-NCI "Common Terminology Criteria for Adverse Events v4.0".
* Pregnant or breast-feeding women.
* History of somatic or psychiatric disease/condition that may interfere with the objectives and assessments of the study.
* Clinically significant illness or clinically relevant trauma within 2 weeks before the administration of the investigational product.
* Current history of malignancy; patients with a secondary tumor in remission of > 5 years can be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- University Hospital Basel, Basel, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This open-label, micro-dosing study with 2 sequentially ascending single peptide doses was conducted in a single study center in Switzerland between 23 June 2014 and 14 January 2015.
Pre-assignment Details: A total of 12 participants with histologically confirmed gastro-entero-pancreatic neuroendocrine tumors (GEP NET) and a previously performed somatostatin receptor scan were treated in this study. Each participant underwent a screening visit within 28 days prior to receiving the study's investigational product (IP).
Groups:
- All Participants: Participants received a single dose of the OPS202 peptide (15 [± 5] microgram (μg) on Day 0. All doses were labeled with 68Ga at a fixed dose of 200 megabecquerel (MBq) (± 25%) per injection. 68Ga-OPS202 was administered intravenously over a time period of less than 1 minute prior to three dimensional (3D) positron emission tomography/computed tomography (PET/CT) scan. As per the sequential dosing scheme, on Day 21, participants then received a single dose of 50 (± 15) μg of 68Ga-OPS202 prior to 3D PET/CT.
Period: Overall Study
Arm/Group | All Participants
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF) included all participants of the full analysis set (FAS) who received the IP, regardless of any protocol deviations.
Groups:
- All Participants: Participants received a single dose of the OPS202 peptide (15 [± 5] μg on Day 0. All doses were labeled with 68Ga at a fixed dose of 200 MBq (± 25%) per injection. 68Ga-OPS202 was administered intravenously over a time period of less than 1 minute prior to 3D PET/CT scan. As per the sequential dosing scheme, on Day 21, participants then received a single dose of 50 (± 15) μg of 68Ga-OPS202 prior to 3D PET/CT.
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (14.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reported With Adverse Events (AEs), Serious Adverse Events (SAEs), and Adverse Drug Reactions (ADRs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a IP and which does not necessarily have a causal relationship with this treatment. For this study, all AEs were regarded as 'treatment emergent', i.e., not seen before administration of the IP or, if already present before administration, worsened after start of administration. An SAE was defined as an event that led to death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect. An ADR was defined as an AE with probable, possible or unlikely relationship to the administration of 68Ga-OPS202.
Time Frame: From start of IP administration to end of the study visit (approximately 28 to 36 days)
Population: The SAF included all participants of the FAS who received the IP, regardless of any protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 12
Participants
  Any AE | 6
  SAEs | 0
  ADRs | 5

2. Primary Outcome: Number of Participants With Clinical Significant Abnormalities in Laboratory Parameters, Vital Signs, Cardiac Safety, Physical Examination, and Required Concomitant Medication
Description: Laboratory assessments included hematology, blood biochemistry and urine analysis. Vital signs included systolic and diastolic blood pressure, heart rate and axillary body temperature. Cardiac safety was assessed by 12-lead ECGs and physical examination included general appearance, head, neck, eyes, ears, nose, throat, respiratory, cardiovascular, gastrointestinal, musculoskeletal, neurological, endocrine, lymphatic, dermatological, psychological/psychiatric, abdomen, and genitourinary body systems. All medications (including herbal products) taken from visit 1 (Day 0) to visit 3 (7-15 days after visit 2 (3-4 weeks after visit 1), end of the study) were recorded in the participant's case report form.
Time Frame: From start of IP administration to end of the study visit (approximately 28 to 36 days)
Population: The SAF included all participants of the FAS who received the investigational product, regardless of any protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 12
Participants
  Laboratory parameters abnormalities | 8
  Vital sign abnormalities | 7
  12-Lead ECG abnormalities | 1
  Physical examination abnormalities | 9
  Concomitant medications required | 12

3. Secondary Outcome: Number of Malignant and Benign Lesions Detected for Session 1
Description: At visit 1, after administration of 15 μg 68Ga-OPS202, a dynamic scan was performed in kidney region over first 30 minutes; static scans were performed from head to sub-inguinal region at 0.5, 1, 2 and 4 h post-injection. At visit 2, after administration of 50 μg 68Ga-OPS202, a static scan was performed from head to sub-inguinal region at 1 h post-injection. A previous somatostatin receptor scan had been performed within 6 months prior to Day 0. Lesions were classified into malignant and benign by readers. Lesion matching was performed between somatostatin receptor scan and 1 h-68Ga-OPS202 receptor scans at visit 1 and visit 2. Number of lesions for each organ/tissue and overall were calculated and absolute numbers reported. Two different read sessions were held to generate data sets for evaluation of target variables. Statistical comparisons were only feasible for those organs/ tissues that had sufficient participants with lesions detected.
Time Frame: 6 months prior to Day 0; and 1 hour post-injection on Day 0 and Day 21
Population: The Intention-to-Treat (ITT) set included all participants of the FAS who received the IP and had at least 1 evaluable PET/CT scan image available for at least 1 time point at visit 1 (Day 0) or visit 2 (Day 21), regardless of any protocol deviations.
Measure: Mean (Standard Deviation); unit: lesion
Groups:
- ITT Population (Pre-dose): Participants had a somatostatin receptor scan performed within 6 months prior to the first injection of IP.
- ITT Population (Day 0): Participants received a single intravenous dose of 15 (± 5) μg of OPS202 peptide plus 68Ga at a fixed dose of 200 MBq (± 25%) per injection on Day 0 prior to PET/CT scan.
- ITT Population (Day 21): Participants received a single intravenous dose of 50 (± 5) μg of OPS202 peptide plus 68Ga at a fixed dose of 200 MBq (± 25%) per injection on Day 21 prior to PET/CT scan.
Arm/Group | ITT Population (Pre-dose) | ITT Population (Day 0) | ITT Population (Day 21)
Number analyzed (Participants) | 12 | 12 | 12
lesion
  Malignant: Total: number analyzed (Participants) | 11 | 11 | 11
  Malignant: Total | 9.3 (10.49) | 17.0 (17.31) | 20.1 (20.58)
  Malignant: Bone: number analyzed (Participants) | 2 | 2 | 2
  Malignant: Bone | 1.0 (0.00) | 1.0 (0.00) | 1.0 (0.00)
  Malignant: Liver: number analyzed (Participants) | 9 | 9 | 9
  Malignant: Liver | 8.6 (10.62) | 17.4 (17.98) | 21.7 (20.86)
  Malignant: Lymph node: number analyzed (Participants) | 8 | 8 | 8
  Malignant: Lymph node | 2.5 (2.56) | 2.9 (2.10) | 2.5 (2.27)
  Malignant: Peritoneum: number analyzed (Participants) | 1 | 1 | 1
  Malignant: Peritoneum | 1.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 1.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 1.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Malignant: Small bowel: number analyzed (Participants) | 2 | 2 | 2
  Malignant: Small bowel | 1.0 (0.00) | 2.0 (1.41) | 1.5 (0.71)
  Benign: Total: number analyzed (Participants) | 4 | 4 | 4
  Benign: Total | 3.0 (1.83) | 1.8 (2.87) | 3.0 (3.16)
  Benign: Lung: number analyzed (Participants) | 1 | 1 | 1
  Benign: Lung | 0.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 2.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 3.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Benign: Lymph node: number analyzed (Participants) | 1 | 1 | 1
  Benign: Lymph node | 1.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 0.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 0.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Benign: Mamma: number analyzed (Participants) | 1 | 1 | 1
  Benign: Mamma | 2.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 2.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 2.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Benign: Mediastinum: number analyzed (Participants) | 1 | 1 | 1
  Benign: Mediastinum | 1.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 0.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 0.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Benign: Pancreas: number analyzed (Participants) | 1 | 1 | 1
  Benign: Pancreas | 1.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 1.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 1.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Benign: Small bowel: number analyzed (Participants) | 1 | 1 | 1
  Benign: Small bowel | 4.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 0.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 4.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Benign: Spleen: number analyzed (Participants) | 1 | 1 | 1
  Benign: Spleen | 1.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 1.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 1.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Benign: Stomach: number analyzed (Participants) | 1 | 1 | 1
  Benign: Stomach | 1.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 1.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 1.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Benign: Thyroid gland: number analyzed (Participants) | 1 | 1 | 1
  Benign: Thyroid gland | 1.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 0.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 0.0 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
Statistical Analysis 1: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 0); Comparison of malignant lesions in total tissues between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 1 receptor scan (ITT population Day 0) at 1 hour time point; Test type: Other; p = 0.016, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 21); Comparison of malignant lesions in total tissues between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 2 receptor scan (ITT population Day 21) at 1 hour time point; Test type: Other; p = 0.004, Wilcoxon signed rank test
Statistical Analysis 3: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 0); Comparison of malignant lesions in liver between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 1 receptor scan (ITT population Day 0) at 1 hour time point; Test type: Other; p = 0.012, Wilcoxon signed rank test
Statistical Analysis 4: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 21); Comparison of malignant lesions in liver between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 2 receptor scan (ITT population Day 21) at 1 hour time point; Test type: Other; p = 0.004, Wilcoxon signed rank test
Statistical Analysis 5: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 0); Comparison of malignant lesions in lymph node between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 1 receptor scan (ITT population Day 0) at 1 hour time point; Test type: Other; p = 0.500, Wilcoxon signed rank test
Statistical Analysis 6: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 21); Comparison of malignant lesions in lymph node between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 2 receptor scan (ITT population Day 21) at 1 hour time point; Test type: Other; p = 1.000, Wilcoxon signed rank test

4. Secondary Outcome: Percentage of Participants With Lesion-Associated 68Ga-OPS202 Binding
Description: Tumor contrast in PET imaging was determined by qualitative visual analysis. 68Ga-OPS202 binding was present if at least one lesion, regardless of nature, was detected within respective tissue location. Percentages were based on number of participants with available scan at corresponding time point.
Time Frame: At 0.5, 1, 2, and 4 hour post-injection on Day 0 and 1 hour post-injection on Day 21
Population: The ITT set included all participants of the FAS who received the IP and had at least 1 evaluable PET/CT scan image available for at least 1 time point at visit 1 (Day 0) or visit 2 (Day 21), regardless of any protocol deviations.
Measure: Number; unit: percentage of participants
Arm/Group | ITT Population (Day 0) | ITT Population (Day 21)
Number analyzed (Participants) | 12 | 12
percentage of participants
  Total: At 0.5 hour: number analyzed (Participants) | 12 | 0
  Total: At 0.5 hour | 100 |
  Total: At 1 hour | 100 | 100
  Total: At 2 hour: number analyzed (Participants) | 12 | 0
  Total: At 2 hour | 100 |
  Total: At 4 hour: number analyzed (Participants) | 12 | 0
  Total: At 4 hour | 100 |
  Bone: At 0.5 hour: number analyzed (Participants) | 12 | 0
  Bone: At 0.5 hour | 16.7 |
  Bone: At 1 hour | 16.7 | 16.7
  Bone: At 2 hour: number analyzed (Participants) | 12 | 0
  Bone: At 2 hour | 16.7 |
  Bone: At 4 hour: number analyzed (Participants) | 12 | 0
  Bone: At 4 hour | 16.7 |
  Liver: At 0.5 hour: number analyzed (Participants) | 12 | 0
  Liver: At 0.5 hour | 75.0 |
  Liver: At 1 hour | 75.0 | 75.0
  Liver: At 2 hour: number analyzed (Participants) | 12 | 0
  Liver: At 2 hour | 75.0 |
  Liver: At 4 hour: number analyzed (Participants) | 12 | 0
  Liver: At 4 hour | 75.0 |
  Lung: At 0.5 hour: number analyzed (Participants) | 12 | 0
  Lung: At 0.5 hour | 0 |
  Lung: At 1 hour | 0 | 0
  Lung: At 2 hour: number analyzed (Participants) | 12 | 0
  Lung: At 2 hour | 0 |
  Lung: At 4 hour: number analyzed (Participants) | 12 | 0
  Lung: At 4 hour | 0 |
  Lymph node: At 0.5 hour: number analyzed (Participants) | 12 | 0
  Lymph node: At 0.5 hour | 58.3 |
  Lymph node: At 1 hour | 58.3 | 58.3
  Lymph node: At 2 hour: number analyzed (Participants) | 12 | 0
  Lymph node: At 2 hour | 58.3 |
  Lymph node: At 4 hour: number analyzed (Participants) | 12 | 0
  Lymph node: At 4 hour | 58.3 |
  Mamma: At 0.5 hour: number analyzed (Participants) | 12 | 0
  Mamma: At 0.5 hour | 0 |
  Mamma: At 1 hour | 0 | 0
  Mamma: At 2 hour: number analyzed (Participants) | 12 | 0
  Mamma: At 2 hour | 0 |
  Mamma: At 4 hour: number analyzed (Participants) | 12 | 0
  Mamma: At 4 hour | 0 |
  Pancreas: At 0.5 hour: number analyzed (Participants) | 12 | 0
  Pancreas: At 0.5 hour | 8.3 |
  Pancreas: At 1 hour | 8.3 | 8.3
  Pancreas: At 2 hour: number analyzed (Participants) | 12 | 0
  Pancreas: At 2 hour | 8.3 |
  Pancreas: At 4 hour: number analyzed (Participants) | 12 | 0
  Pancreas: At 4 hour | 8.3 |
  Peritoneum: At 0.5 hour: number analyzed (Participants) | 12 | 0
  Peritoneum: At 0.5 hour | 8.3 |
  Peritoneum: At 1 hour | 8.3 | 8.3
  Peritoneum: At 2 hour: number analyzed (Participants) | 12 | 0
  Peritoneum: At 2 hour | 8.3 |
  Peritoneum: At 4 hour: number analyzed (Participants) | 12 | 0
  Peritoneum: At 4 hour | 8.3 |
  Small bowel: At 0.5 hour: number analyzed (Participants) | 12 | 0
  Small bowel: At 0.5 hour | 25.0 |
  Small bowel: At 1 hour | 25.0 | 25.0
  Small bowel: At 2 hour: number analyzed (Participants) | 12 | 0
  Small bowel: At 2 hour | 25.0 |
  Small bowel: At 4 hour: number analyzed (Participants) | 12 | 0
  Small bowel: At 4 hour | 16.7 |
  Thyroid gland: At 0.5 hour: number analyzed (Participants) | 12 | 0
  Thyroid gland: At 0.5 hour | 0 |
  Thyroid gland: At 1 hour | 0 | 0
  Thyroid gland: At 2 hour: number analyzed (Participants) | 12 | 0
  Thyroid gland: At 2 hour | 0 |
  Thyroid gland: At 4 hour: number analyzed (Participants) | 12 | 0
  Thyroid gland: At 4 hour | 0 |

5. Secondary Outcome: Mean Maximum Standardized Uptake Value (SUVmax) of Malignant and Benign Lesions for Session 1
Description: At visit 1, after administration of 15 μg 68Ga-OPS202, a dynamic scan was performed in kidney region over the first 30 minutes (0-0.5 h); static scans were performed from head to sub-inguinal region at 0.5, 1, 2 and 4 h post-injection. At visit 2, after administration of 50 μg 68Ga-OPS202, a static scan was performed from head to sub-inguinal region at 1 h post-injection. A previous somatostatin receptor scan had been performed within 6 months prior to Day 0. Lesions were classified into malignant and benign lesion by the readers according to their experience. Lesion matching was performed between the somatostatin receptor scan and the 1 h-68Ga-OPS202 receptor scans at visit 1 and visit 2. The mean SUVmax of lesions (mean of all identified lesions in the lymph node and liver) was summarized by nature of the lesions (malignant, benign). Statistical comparisons were only feasible for those organs/ tissues that had sufficient participants with lesions detected.
Time Frame: 6 months prior to Day 0; and 1 hour post-injection on Day 0 and Day 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: SUVmax
Arm/Group | ITT Population (Pre-dose) | ITT Population (Day 0) | ITT Population (Day 21)
Number analyzed (Participants) | 12 | 12 | 12
SUVmax
  Malignant: Bone: number analyzed (Participants) | 2 | 2 | 2
  Malignant: Bone | 4.394 (0.9396) | 4.153 (2.0270) | 4.455 (0.2425)
  Malignant: Liver: number analyzed (Participants) | 9 | 9 | 9
  Malignant: Liver | 12.135 (4.4660) | 10.468 (4.7970) | 8.458 (3.4840)
  Malignant: Lymph node: number analyzed (Participants) | 7 | 8 | 8
  Malignant: Lymph node | 15.192 (7.4318) | 16.289 (12.0091) | 14.602 (10.9725)
  Malignant: Peritoneum: number analyzed (Participants) | 1 | 1 | 1
  Malignant: Peritoneum | 6.579 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 6.740 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 9.504 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Malignant: Small bowel: number analyzed (Participants) | 2 | 2 | 2
  Malignant: Small bowel | 14.049 (0.2124) | 11.140 (7.9828) | 9.156 (1.0674)
  Benign: Lung: number analyzed (Participants) | 0 | 1 | 1
  Benign: Lung |  | 3.410 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 3.131 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Benign: Lymph node: number analyzed (Participants) | 1 | 0 | 0
  Benign: Lymph node | 3.093 (NA) — Standard deviation cannot be calculated when only one participant analyzed. |  |
  Benign: Mamma: number analyzed (Participants) | 1 | 1 | 1
  Benign: Mamma | 2.353 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 2.907 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 2.538 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Benign: Mediastinum: number analyzed (Participants) | 1 | 0 | 0
  Benign: Mediastinum | 2.242 (NA) — Standard deviation cannot be calculated when only one participant analyzed. |  |
  Benign: Pancreas: number analyzed (Participants) | 1 | 1 | 1
  Benign: Pancreas | 14.086 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 8.693 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 6.659 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Benign: Small bowel: number analyzed (Participants) | 1 | 0 | 1
  Benign: Small bowel | 8.264 (NA) — Standard deviation cannot be calculated when only one participant analyzed. |  | 4.990 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Benign: Spleen: number analyzed (Participants) | 1 | 1 | 1
  Benign: Spleen | 16.343 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 15.997 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 14.308 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Benign: Stomach: number analyzed (Participants) | 1 | 1 | 1
  Benign: Stomach | 6.713 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 7.630 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 5.305 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Benign: Thyroid gland: number analyzed (Participants) | 1 | 0 | 0
  Benign: Thyroid gland | 3.768 (NA) — Standard deviation cannot be calculated when only one participant analyzed. |  |
Statistical Analysis 1: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 0); Comparison of SUVmax of malignant lesions in liver between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 1 receptor scan (ITT population Day 0) at 1 hour time point; Test type: Other; p = 0.250, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 21); Comparison of SUVmax of malignant lesions in liver between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 2 receptor scan (ITT population Day 21) at 1 hour time point; Test type: Other; p = 0.004, Wilcoxon signed rank test
Statistical Analysis 3: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 0); Comparison of SUVmax of malignant lesions in lymph node between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 1 receptor scan (ITT population Day 0) at 1 hour time point; Test type: Other; p = 0.688, Wilcoxon signed rank test
Statistical Analysis 4: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 21); Comparison of SUVmax of malignant lesions in lymph node between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 2 receptor scan (ITT population Day 21) at 1 hour time point; Test type: Other; p = 0.578, Wilcoxon signed rank test

6. Secondary Outcome: Mean SUVmax of Malignant and Benign Lesions for Session 2
Description: The mean SUVmax of all identified lesions in the respective organ/tissue was determined. Statistical comparisons were only feasible for those organs/ tissues that had sufficient participants with lesions detected.
Time Frame: At 0.5, 1, 2, and 4 hour post-injection on Day 0 and 1 hour post-injection on Day 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: SUVmax
Arm/Group | ITT Population (Day 0) | ITT Population (Day 21)
Number analyzed (Participants) | 12 | 12
SUVmax
  Malignant: Bone: At 0.5 hour: number analyzed (Participants) | 2 | 0
  Malignant: Bone: At 0.5 hour | 4.938 (1.1179) |
  Malignant: Bone: At 1 hour: number analyzed (Participants) | 2 | 2
  Malignant: Bone: At 1 hour | 4.153 (2.0270) | 4.455 (0.2425)
  Malignant: Bone: At 2 hour: number analyzed (Participants) | 2 | 0
  Malignant: Bone: At 2 hour | 4.601 (1.3164) |
  Malignant: Bone: At 4 hour: number analyzed (Participants) | 2 | 0
  Malignant: Bone: At 4 hour | 4.564 (1.0832) |
  Malignant: Liver: At 0.5 hour: number analyzed (Participants) | 9 | 0
  Malignant: Liver: At 0.5 hour | 10.086 (5.0229) |
  Malignant: Liver: At 1 hour: number analyzed (Participants) | 9 | 9
  Malignant: Liver: At 1 hour | 11.485 (6.3691) | 9.037 (3.9033)
  Malignant: Liver: At 2 hour: number analyzed (Participants) | 9 | 0
  Malignant: Liver: At 2 hour | 9.897 (4.3537) |
  Malignant: Liver: At 4 hour: number analyzed (Participants) | 9 | 0
  Malignant: Liver: At 4 hour | 12.482 (5.9410) |
  Malignant: Lymph node: At 0.5 hour: number analyzed (Participants) | 7 | 0
  Malignant: Lymph node: At 0.5 hour | 14.581 (9.7609) |
  Malignant: Lymph node: At 1 hour: number analyzed (Participants) | 7 | 7
  Malignant: Lymph node: At 1 hour | 17.044 (11.6224) | 15.836 (10.9868)
  Malignant: Lymph node: At 2 hour: number analyzed (Participants) | 7 | 0
  Malignant: Lymph node: At 2 hour | 18.166 (10.6940) |
  Malignant: Lymph node: At 4 hour: number analyzed (Participants) | 7 | 0
  Malignant: Lymph node: At 4 hour | 17.985 (13.5368) |
  Malignant: Peritoneum: At 0.5 hour: number analyzed (Participants) | 1 | 0
  Malignant: Peritoneum: At 0.5 hour | 3.293 (NA) — Standard deviation cannot be calculated when only one participant analyzed. |
  Malignant: Peritoneum: At 1 hour: number analyzed (Participants) | 1 | 1
  Malignant: Peritoneum: At 1 hour | 6.740 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 9.504 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Malignant: Peritoneum: At 2 hour: number analyzed (Participants) | 1 | 0
  Malignant: Peritoneum: At 2 hour | 7.484 (NA) — Standard deviation cannot be calculated when only one participant analyzed. |
  Malignant: Peritoneum: At 4 hour: number analyzed (Participants) | 1 | 0
  Malignant: Peritoneum: At 4 hour | 7.216 (NA) — Standard deviation cannot be calculated when only one participant analyzed. |
  Malignant: Small bowel: At 0.5 hour: number analyzed (Participants) | 3 | 0
  Malignant: Small bowel: At 0.5 hour | 9.474 (5.8641) |
  Malignant: Small bowel: At 1 hour: number analyzed (Participants) | 3 | 3
  Malignant: Small bowel: At 1 hour | 11.207 (4.5367) | 7.440 (2.8588)
  Malignant: Small bowel: At 2 hour: number analyzed (Participants) | 3 | 0
  Malignant: Small bowel: At 2 hour | 9.075 (4.9059) |
  Malignant: Small bowel: At 4 hour: number analyzed (Participants) | 2 | 0
  Malignant: Small bowel: At 4 hour | 14.695 (6.9926) |
  Benign: Pancreas: At 0.5 hour: number analyzed (Participants) | 1 | 0
  Benign: Pancreas: At 0.5 hour | 8.561 (NA) — Standard deviation cannot be calculated when only one participant analyzed. |
  Benign: Pancreas: At 1 hour: number analyzed (Participants) | 1 | 1
  Benign: Pancreas: At 1 hour | 8.512 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 6.659 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Benign: Pancreas: At 2 hour: number analyzed (Participants) | 1 | 0
  Benign: Pancreas: At 2 hour | 8.734 (NA) — Standard deviation cannot be calculated when only one participant analyzed. |
  Benign: Pancreas: At 4 hour: number analyzed (Participants) | 1 | 0
  Benign: Pancreas: At 4 hour | 5.759 (NA) — Standard deviation cannot be calculated when only one participant analyzed. |
Statistical Analysis 1: Comparison: ITT Population (Day 0) vs ITT Population (Day 21); Comparison of SUVmax of malignant lesions in liver between 68Ga-OPS202 visit 1 receptor scan (ITT population Day 0) and the 68Ga-OPS202 visit 2 receptor scan (ITT population Day 21) at 1 hour time point; Test type: Other; p = 0.027, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: ITT Population (Day 0) vs ITT Population (Day 21); Comparison of SUVmax of malignant lesions in lymph node between 68Ga-OPS202 visit 1 receptor scan (ITT population Day 0) and the 68Ga-OPS202 visit 2 receptor scan (ITT population Day 21) at 1 hour time point; Test type: Other; p = 0.219, Wilcoxon signed rank test

7. Secondary Outcome: Mean SUVmax of Reference Tissues (RT) Region of Interests (ROIs) for Session 1
Description: Lesion matching was performed between somatostatin receptor scan and 1 h-68Ga-OPS202 receptor scans at visit 1 and visit 2. Mean SUVmax of all selected ROIs in corresponding RT was determined. Corresponding RTs were adjacent healthy regions (1 to 3 healthy regions were identified for each lesion), i.e. located in same organ and/or region as lesion. RTs were determined in tissue locations with malignant lesions only. ROIs were also selected in muscle tissue, which was used as an additional reference region. Statistical comparisons were only feasible for those organs/ tissues that had sufficient participants with lesions detected.
Time Frame: 6 months prior to Day 0; and 1 hour post-injection on Day 0 and Day 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: SUVmax
Arm/Group | ITT Population (Pre-dose) | ITT Population (Day 0) | ITT Population (Day 21)
Number analyzed (Participants) | 12 | 12 | 12
SUVmax
  Bone: number analyzed (Participants) | 2 | 2 | 2
  Bone | 0.610 (0.1801) | 0.739 (0.1780) | 0.636 (0.1207)
  Muscle | 1.020 (0.3141) | 0.883 (0.2530) | 0.896 (0.1812)
  Liver | 6.801 (1.9676) | 3.642 (1.6381) | 2.959 (0.8089)
  Lymph node: number analyzed (Participants) | 7 | 8 | 8
  Lymph node | 2.229 (1.2017) | 1.870 (0.6967) | 2.368 (1.7112)
  Peritoneum: number analyzed (Participants) | 1 | 1 | 1
  Peritoneum | 0.776 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 0.927 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 1.401 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Small bowel: number analyzed (Participants) | 2 | 2 | 2
  Small bowel | 4.180 (0.7893) | 2.080 (0.5162) | 1.707 (0.0636)
Statistical Analysis 1: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 0); Comparison of SUVmax of RT in muscle between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 1 receptor scan (ITT population Day 0) at 1 hour time point; Test type: Other; p = 0.064, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 21); Comparison of SUVmax of RT in muscle between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 2 receptor scan (ITT population Day 21) at 1 hour time point; Test type: Other; p = 0.339, Wilcoxon signed rank test
Statistical Analysis 3: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 0); Comparison of SUVmax of RT in liver between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 1 receptor scan (ITT population Day 0) at 1 hour time point; Test type: Other; p = 0.001, Wilcoxon signed rank test
Statistical Analysis 4: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 21); Comparison of SUVmax of RT in liver between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 2 receptor scan (ITT population Day 21) at 1 hour time point; Test type: Other; p = 0.000, Wilcoxon signed rank test
Statistical Analysis 5: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 0); Comparison of SUVmax of RT in lymph node between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 1 receptor scan (ITT population Day 0) at 1 hour time point; Test type: Other; p = 0.297, Wilcoxon signed rank test
Statistical Analysis 6: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 21); Comparison of SUVmax of RT in lymph node between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 2 receptor scan (ITT population Day 21) at 1 hour time point; Test type: Other; p = 1.000, Wilcoxon signed rank test

8. Secondary Outcome: Mean SUVmax of RT for Session 2
Description: The mean SUVmax of all selected ROIs in the corresponding RT was determined. RTs were determined in tissue locations with malignant lesions only. ROIs were also selected in muscle tissue, which was used as an additional reference region. Statistical comparisons were only feasible for those organs/ tissues that had sufficient participants with lesions detected.
Time Frame: At 0.5, 1, 2, and 4 hour post-injection on Day 0 and 1 hour post-injection on Day 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: SUVmax
Arm/Group | ITT Population (Day 0) | ITT Population (Day 21)
Number analyzed (Participants) | 12 | 12
SUVmax
  Muscle: At 0.5 hour: number analyzed (Participants) | 12 | 0
  Muscle: At 0.5 hour | 0.923 (0.2260) |
  Muscle: At 1 hour | 0.932 (0.2386) | 0.976 (0.2012)
  Muscle: At 2 hour: number analyzed (Participants) | 12 | 0
  Muscle: At 2 hour | 1.127 (0.3343) |
  Muscle: At 4 hour: number analyzed (Participants) | 12 | 0
  Muscle: At 4 hour | 2.013 (0.6884) |
  Bone: At 0.5 hour: number analyzed (Participants) | 2 | 0
  Bone: At 0.5 hour | 0.573 (0.3418) |
  Bone: At 1 hour: number analyzed (Participants) | 2 | 2
  Bone: At 1 hour | 0.605 (0.3681) | 0.765 (0.1409)
  Bone: At 2 hour: number analyzed (Participants) | 2 | 0
  Bone: At 2 hour | 0.731 (0.0550) |
  Bone: At 4 hour: number analyzed (Participants) | 2 | 0
  Bone: At 4 hour | 2.138 (0.7022) |
  Liver: At 0.5 hour: number analyzed (Participants) | 12 | 0
  Liver: At 0.5 hour | 4.201 (1.3697) |
  Liver: At 1 hour | 4.040 (1.5213) | 3.480 (1.1863)
  Liver: At 2 hour: number analyzed (Participants) | 12 | 0
  Liver: At 2 hour | 4.103 (1.2389) |
  Liver: At 4 hour: number analyzed (Participants) | 12 | 0
  Liver: At 4 hour | 6.101 (2.7773) |
  Lymph node: At 0.5 hour: number analyzed (Participants) | 7 | 0
  Lymph node: At 0.5 hour | 1.723 (0.9118) |
  Lymph node: At 1 hour: number analyzed (Participants) | 7 | 7
  Lymph node: At 1 hour | 2.049 (0.7805) | 1.757 (1.1486)
  Lymph node: At 2 hour: number analyzed (Participants) | 7 | 0
  Lymph node: At 2 hour | 2.467 (1.3033) |
  Lymph node: At 4 hour: number analyzed (Participants) | 7 | 0
  Lymph node: At 4 hour | 1.989 (0.6904) |
  Peritoneum: At 0.5 hour: number analyzed (Participants) | 1 | 0
  Peritoneum: At 0.5 hour | 1.864 (NA) — Standard deviation cannot be calculated when only one participant analyzed. |
  Peritoneum: At 1 hour: number analyzed (Participants) | 1 | 1
  Peritoneum: At 1 hour | 1.038 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 1.163 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Peritoneum: At 2 hour: number analyzed (Participants) | 1 | 0
  Peritoneum: At 2 hour | 0.856 (NA) — Standard deviation cannot be calculated when only one participant analyzed. |
  Peritoneum: At 4 hour: number analyzed (Participants) | 1 | 0
  Peritoneum: At 4 hour | 1.501 (NA) — Standard deviation cannot be calculated when only one participant analyzed. |
  Small bowel: At 0.5 hour: number analyzed (Participants) | 3 | 0
  Small bowel: At 0.5 hour | 2.519 (0.2743) |
  Small bowel: At 1 hour: number analyzed (Participants) | 3 | 3
  Small bowel: At 1 hour | 2.571 (1.0644) | 1.608 (0.3677)
  Small bowel: At 2 hour: number analyzed (Participants) | 3 | 0
  Small bowel: At 2 hour | 2.124 (0.7382) |
  Small bowel: At 4 hour: number analyzed (Participants) | 3 | 0
  Small bowel: At 4 hour | 3.177 (0.7174) |
Statistical Analysis 1: Comparison: ITT Population (Day 0) vs ITT Population (Day 21); Comparison of SUVmax of RT in muscle between 68Ga-OPS202 visit 1 receptor scan (ITT population Day 0) and the 68Ga-OPS202 visit 2 receptor scan (ITT population Day 21) at 1 hour time point; Test type: Other; p = 0.470, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: ITT Population (Day 0) vs ITT Population (Day 21); Comparison of SUVmax of RT in liver between 68Ga-OPS202 visit 1 receptor scan (ITT population Day 0) and the 68Ga-OPS202 visit 2 receptor scan (ITT population Day 21) at 1 hour time point; Test type: Other; p = 0.233, Wilcoxon signed rank test
Statistical Analysis 3: Comparison: ITT Population (Day 0) vs ITT Population (Day 21); Comparison of SUVmax of RT in lymph node between 68Ga-OPS202 visit 1 receptor scan (ITT population Day 0) and the 68Ga-OPS202 visit 2 receptor scan (ITT population Day 21) at 1 hour time point; Test type: Other; p = 0.375, Wilcoxon signed rank test

9. Secondary Outcome: Mean Tumor Contrast (3D-SUV-R) of Malignant Lesions Compared to Pre-dose Scans for Session 1
Description: The tumor contrast, i.e. the SUV ratio for tumor (malignant lesion)-to-background (3D-SUV-R) of a single lesion was defined as: 3D-SUV-R = SUVmax of lesion / mean of SUVmax of corresponding RTs. Statistical comparisons were only feasible for those organs/ tissues that had sufficient participants with lesions detected.
Time Frame: 6 months prior to Day 0; and 1 hour post-injection on Day 0 and Day 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ITT Population (Pre-dose) | ITT Population (Day 0) | ITT Population (Day 21)
Number analyzed (Participants) | 12 | 12 | 12
ratio
  Bone (RT: Bone): number analyzed (Participants) | 2 | 2 | 2
  Bone (RT: Bone) | 7.296 (0.6136) | 6.125 (4.2161) | 7.167 (1.7409)
  Bone (RT: Muscle): number analyzed (Participants) | 2 | 2 | 2
  Bone (RT: Muscle) | 5.227 (1.7044) | 6.091 (2.1353) | 5.868 (0.4515)
  Liver (RT: Liver): number analyzed (Participants) | 9 | 9 | 9
  Liver (RT: Liver) | 2.066 (0.9163) | 3.234 (1.8130) | 3.215 (1.8160)
  Liver (RT: Muscle): number analyzed (Participants) | 9 | 9 | 9
  Liver (RT: Muscle) | 13.434 (7.3703) | 12.605 (7.9383) | 10.318 (5.7811)
  Lymph node (RT: Lymph node): number analyzed (Participants) | 7 | 8 | 8
  Lymph node (RT: Lymph node) | 9.548 (7.1592) | 9.320 (5.2590) | 11.034 (13.3938)
  Lymph node (RT: Muscle): number analyzed (Participants) | 7 | 8 | 8
  Lymph node (RT: Muscle) | 15.110 (7.4282) | 19.861 (16.0492) | 18.349 (15.9027)
  Peritoneum (RT: Peritoneum): number analyzed (Participants) | 1 | 1 | 1
  Peritoneum (RT: Peritoneum) | 8.475 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 7.268 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 6.783 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Peritoneum (RT: Muscle): number analyzed (Participants) | 1 | 1 | 1
  Peritoneum (RT: Muscle) | 8.366 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 9.170 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 11.399 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Small bowel (RT: Small bowel): number analyzed (Participants) | 2 | 2 | 2
  Small bowel (RT: Small bowel) | 3.427 (0.6978) | 6.017 (5.3303) | 5.355 (0.4256)
  Small bowel (RT: Muscle): number analyzed (Participants) | 2 | 2 | 2
  Small bowel (RT: Muscle) | 15.353 (7.1430) | 12.585 (6.1981) | 11.352 (2.5753)
Statistical Analysis 1: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 0); Comparison of 3D-SUV-R of malignant lesions in liver with RT as liver between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 1 receptor scan (ITT population Day 0) at 1 hour time point; Test type: Other; p = 0.004, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 21); Comparison of 3D-SUV-R of malignant lesions in liver with RT as liver between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 2 receptor scan (ITT population Day 21) at 1 hour time point; Test type: Other; p = 0.004, Wilcoxon signed rank test
Statistical Analysis 3: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 0); Comparison of 3D-SUV-R of malignant lesions in liver with RT as muscle between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 1 receptor scan (ITT population Day 0) at 1 hour time point; Test type: Other; p = 0.426, Wilcoxon signed rank test
Statistical Analysis 4: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 21); Comparison of 3D-SUV-R of malignant lesions in liver with RT as muscle between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 2 receptor scan (ITT population Day 21) at 1 hour time point; Test type: Other; p = 0.098, Wilcoxon signed rank test
Statistical Analysis 5: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 0); Comparison of 3D-SUV-R of malignant lesions in lymph node with RT as lymph node between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 1 receptor scan (ITT population Day 0) at 1 hour time point; Test type: Other; p = 0.813, Wilcoxon signed rank test
Statistical Analysis 6: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 21); Comparison of 3D-SUV-R of malignant lesions in lymph node with RT as lymph node between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 2 receptor scan (ITT population Day 21) at 1 hour time point; Test type: Other; p = 0.813, Wilcoxon signed rank test
Statistical Analysis 7: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 0); Comparison of 3D-SUV-R of malignant lesions in lymph node with RT as muscle between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 1 receptor scan (ITT population Day 0) at 1 hour time point; Test type: Other; p = 0.297, Wilcoxon signed rank test
Statistical Analysis 8: Comparison: ITT Population (Pre-dose) vs ITT Population (Day 21); Comparison of 3D-SUV-R of malignant lesions in lymph node with RT as muscle between previous somatostatin receptor scan (ITT population pre-dose) and the 68Ga-OPS202 visit 2 receptor scan (ITT population Day 21) at 1 hour time point; Test type: Other; p = 0.469, Wilcoxon signed rank test

10. Secondary Outcome: The 3D-SUV-R of Malignant Lesions for Session 2
Description: The tumor contrast, i.e. the SUV ratio for 3D-SUV-R of a single lesion was defined as: 3D-SUV-R = SUVmax of lesion / mean of SUVmax of corresponding RTs. Statistical comparisons were only feasible for those organs/ tissues that had sufficient participants with lesions detected.
Time Frame: At 0.5, 1, 2, and 4 hour post-injection on Day 0 and 1 hour post-injection on Day 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ITT Population (Day 0) | ITT Population (Day 21)
Number analyzed (Participants) | 12 | 12
ratio
  Bone (RT: Bone): At 0.5 hour: number analyzed (Participants) | 2 | 0
  Bone (RT: Bone): At 0.5 hour | 11.191 (8.6266) |
  Bone (RT: Bone): At 1 hour: number analyzed (Participants) | 2 | 2
  Bone (RT: Bone): At 1 hour | 9.679 (9.2426) | 5.891 (0.7682)
  Bone (RT: Bone): At 2 hour: number analyzed (Participants) | 2 | 0
  Bone (RT: Bone): At 2 hour | 6.243 (1.3313) |
  Bone (RT: Bone): At 4 hour: number analyzed (Participants) | 2 | 0
  Bone (RT: Bone): At 4 hour | 2.169 (0.2056) |
  Bone (RT: Muscle): At 0.5 hour: number analyzed (Participants) | 2 | 0
  Bone (RT: Muscle): At 0.5 hour | 6.716 (1.4013) |
  Bone (RT: Muscle): At 1 hour: number analyzed (Participants) | 2 | 2
  Bone (RT: Muscle): At 1 hour | 5.528 (2.1555) | 5.530 (0.8944)
  Bone (RT: Muscle): At 2 hour: number analyzed (Participants) | 2 | 0
  Bone (RT: Muscle): At 2 hour | 5.311 (2.1658) |
  Bone (RT: Muscle): At 4 hour: number analyzed (Participants) | 2 | 0
  Bone (RT: Muscle): At 4 hour | 2.331 (0.5535) |
  Liver (RT: Liver): At 0.5 hour: number analyzed (Participants) | 9 | 0
  Liver (RT: Liver): At 0.5 hour | 2.547 (1.5468) |
  Liver (RT: Liver): At 1 hour: number analyzed (Participants) | 9 | 9
  Liver (RT: Liver): At 1 hour | 3.071 (2.3858) | 2.514 (0.6087)
  Liver (RT: Liver): At 2 hour: number analyzed (Participants) | 9 | 0
  Liver (RT: Liver): At 2 hour | 2.430 (0.9559) |
  Liver (RT: Liver): At 4 hour: number analyzed (Participants) | 9 | 0
  Liver (RT: Liver): At 4 hour | 2.038 (0.6822) |
  Liver (RT: Muscle): At 0.5 hour: number analyzed (Participants) | 9 | 0
  Liver (RT: Muscle): At 0.5 hour | 11.534 (8.0671) |
  Liver (RT: Muscle): At 1 hour: number analyzed (Participants) | 9 | 9
  Liver (RT: Muscle): At 1 hour | 13.231 (10.4892) | 9.653 (5.1879)
  Liver (RT: Muscle): At 2 hour: number analyzed (Participants) | 9 | 0
  Liver (RT: Muscle): At 2 hour | 9.383 (6.1356) |
  Liver (RT: Muscle): At 4 hour: number analyzed (Participants) | 9 | 0
  Liver (RT: Muscle): At 4 hour | 6.974 (6.4729) |
  Lymph node (RT: Lymph node): At 0.5 hour: number analyzed (Participants) | 7 | 0
  Lymph node (RT: Lymph node): At 0.5 hour | 13.448 (12.3973) |
  Lymph node (RT: Lymph node): At 1 hour: number analyzed (Participants) | 7 | 7
  Lymph node (RT: Lymph node): At 1 hour | 10.109 (7.3722) | 14.166 (13.4067)
  Lymph node (RT: Lymph node): At 2 hour: number analyzed (Participants) | 7 | 0
  Lymph node (RT: Lymph node): At 2 hour | 9.722 (7.1821) |
  Lymph node (RT: Lymph node): At 4 hour: number analyzed (Participants) | 7 | 0
  Lymph node (RT: Lymph node): At 4 hour | 9.889 (5.8842) |
  Lymph node (RT: Muscle): At 0.5 hour: number analyzed (Participants) | 7 | 0
  Lymph node (RT: Muscle): At 0.5 hour | 16.362 (9.1362) |
  Lymph node (RT: Muscle): At 1 hour: number analyzed (Participants) | 7 | 7
  Lymph node (RT: Muscle): At 1 hour | 20.434 (13.6060) | 18.562 (15.1302)
  Lymph node (RT: Muscle): At 2 hour: number analyzed (Participants) | 7 | 0
  Lymph node (RT: Muscle): At 2 hour | 16.107 (9.5271) |
  Lymph node (RT: Muscle): At 4 hour: number analyzed (Participants) | 7 | 0
  Lymph node (RT: Muscle): At 4 hour | 8.619 (3.7444) |
  Peritoneum (RT: Peritoneum): At 0.5 hour: number analyzed (Participants) | 1 | 0
  Peritoneum (RT: Peritoneum): At 0.5 hour | 1.767 (NA) — Standard deviation cannot be calculated when only one participant analyzed. |
  Peritoneum (RT: Peritoneum): At 1 hour: number analyzed (Participants) | 1 | 1
  Peritoneum (RT: Peritoneum): At 1 hour | 6.494 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 8.173 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Peritoneum (RT: Peritoneum): At 2 hour: number analyzed (Participants) | 1 | 0
  Peritoneum (RT: Peritoneum): At 2 hour | 8.747 (NA) — Standard deviation cannot be calculated when only one participant analyzed. |
  Peritoneum (RT: Peritoneum): At 4 hour: number analyzed (Participants) | 1 | 0
  Peritoneum (RT: Peritoneum): At 4 hour | 4.809 (NA) — Standard deviation cannot be calculated when only one participant analyzed. |
  Peritoneum (RT: Muscle): At 0.5 hour: number analyzed (Participants) | 1 | 0
  Peritoneum (RT: Muscle): At 0.5 hour | 4.431 (NA) — Standard deviation cannot be calculated when only one participant analyzed. |
  Peritoneum (RT: Muscle): At 1 hour: number analyzed (Participants) | 1 | 1
  Peritoneum (RT: Muscle): At 1 hour | 8.508 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 10.060 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Peritoneum (RT: Muscle): At 2 hour: number analyzed (Participants) | 1 | 0
  Peritoneum (RT: Muscle): At 2 hour | 7.709 (NA) — Standard deviation cannot be calculated when only one participant analyzed. |
  Peritoneum (RT: Muscle): At 4 hour: number analyzed (Participants) | 1 | 0
  Peritoneum (RT: Muscle): At 4 hour | 2.626 (NA) — Standard deviation cannot be calculated when only one participant analyzed. |
  Small bowel (RT: Small bowel): At 0.5 hour: number analyzed (Participants) | 3 | 0
  Small bowel (RT: Small bowel): At 0.5 hour | 3.759 (2.1690) |
  Small bowel (RT: Small bowel): At 1 hour: number analyzed (Participants) | 3 | 3
  Small bowel (RT: Small bowel): At 1 hour | 5.644 (4.9619) | 4.956 (2.8311)
  Small bowel (RT: Small bowel): At 2 hour: number analyzed (Participants) | 3 | 0
  Small bowel (RT: Small bowel): At 2 hour | 4.363 (2.5614) |
  Small bowel (RT: Small bowel): At 4 hour: number analyzed (Participants) | 2 | 0
  Small bowel (RT: Small bowel): At 4 hour | 4.047 (1.6457) |
  Small bowel (RT: Muscle): At 0.5 hour: number analyzed (Participants) | 3 | 0
  Small bowel (RT: Muscle): At 0.5 hour | 9.404 (5.2820) |
  Small bowel (RT: Muscle): At 1 hour: number analyzed (Participants) | 3 | 3
  Small bowel (RT: Muscle): At 1 hour | 11.787 (5.8090) | 7.678 (3.9023)
  Small bowel (RT: Muscle): At 2 hour: number analyzed (Participants) | 3 | 0
  Small bowel (RT: Muscle): At 2 hour | 7.267 (3.8995) |
  Small bowel (RT: Muscle): At 4 hour: number analyzed (Participants) | 2 | 0
  Small bowel (RT: Muscle): At 4 hour | 6.686 (1.5046) |
Statistical Analysis 1: Comparison: ITT Population (Day 0) vs ITT Population (Day 21); Comparison of 3D-SUV-R of malignant lesions in liver with RT as liver between 68Ga-OPS202 visit 1 receptor scan (ITT population Day 0) and 68Ga-OPS202 visit 2 receptor scan (ITT population Day 21) at 1 hour time point; Test type: Other; p = 0.910, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: ITT Population (Day 0) vs ITT Population (Day 21); Comparison of 3D-SUV-R of malignant lesions in liver with RT as muscle between 68Ga-OPS202 visit 1 receptor scan (ITT population Day 0) and 68Ga-OPS202 visit 2 receptor scan (ITT population Day 21) at 1 hour time point; Test type: Other; p = 0.039, Wilcoxon signed rank test
Statistical Analysis 3: Comparison: ITT Population (Day 0) vs ITT Population (Day 21); Comparison of 3D-SUV-R of malignant lesions in lymph node with RT as lymph node between 68Ga-OPS202 visit 1 receptor scan (ITT population Day 0) and 68Ga-OPS202 visit 2 receptor scan (ITT population Day 21) at 1 hour time point; Test type: Other; p = 0.375, Wilcoxon signed rank test
Statistical Analysis 4: Comparison: ITT Population (Day 0) vs ITT Population (Day 21); Comparison of 3D-SUV-R of malignant lesions in lymph node with RT as muscle between 68Ga-OPS202 visit 1 receptor scan (ITT population Day 0) and 68Ga-OPS202 visit 2 receptor scan (ITT population Day 21) at 1 hour time point; Test type: Other; p = 0.219, Wilcoxon signed rank test

11. Secondary Outcome: Percent Change in 3D-SUV-R of Malignant Lesions
Description: The tumor contrast, i.e. the SUV ratio for 3D-SUV-R of a single lesion was defined as: 3D-SUV-R = SUVmax of lesion / mean of SUVmax of corresponding RT. For percent change, 68Ga-OPS202 receptor scan is compared to previous somatostatin receptor scan.
Time Frame: 6 months prior to Day 0; and 1 hour post-injection on Day 0 and Day 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ITT Population (Day 0) | ITT Population (Day 21)
Number analyzed (Participants) | 12 | 12
percent change
  Bone (RT: Bone): number analyzed (Participants) | 2 | 2
  Bone (RT: Bone) | -13.315 (65.0759) | -0.418 (32.2352)
  Bone (RT: Muscle): number analyzed (Participants) | 2 | 2
  Bone (RT: Muscle) | 16.042 (3.0132) | 20.052 (47.7825)
  Liver (RT: Liver): number analyzed (Participants) | 9 | 9
  Liver (RT: Liver) | 51.938 (33.2221) | 50.766 (25.4179)
  Liver (RT: Muscle): number analyzed (Participants) | 9 | 9
  Liver (RT: Muscle) | -5.165 (32.3975) | -19.838 (37.5669)
  Lymph node (RT: Lymph node): number analyzed (Participants) | 7 | 7
  Lymph node (RT: Lymph node) | 56.044 (94.8768) | 38.530 (117.3139)
  Lymph node (RT: Muscle): number analyzed (Participants) | 7 | 7
  Lymph node (RT: Muscle) | 46.569 (61.4515) | 36.864 (79.3287)
  Peritoneum (RT: Peritoneum): number analyzed (Participants) | 1 | 1
  Peritoneum (RT: Peritoneum) | -14.239 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | -19.962 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Peritoneum (RT: Muscle): number analyzed (Participants) | 1 | 1
  Peritoneum (RT: Muscle) | 9.619 (NA) — Standard deviation cannot be calculated when only one participant analyzed. | 36.256 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Small bowel (RT: Small bowel): number analyzed (Participants) | 2 | 2
  Small bowel (RT: Small bowel) | 63.131 (122.3379) | 58.296 (19.8143)
  Small bowel (RT: Muscle): number analyzed (Participants) | 2 | 2
  Small bowel (RT: Muscle) | 2.447 (88.0324) | -12.716 (57.3817)

12. Secondary Outcome: Number of Participants at Each Time Point With the Highest Observed Lesion Number Per Tissue Location
Description: For determining a suitable time window for PET/CT with 68Ga-OPS202, the scans after administration of the 15 μg peptide dose were analyzed and the time point with the highest lesion number per tissue location and overall were determined. If the highest number of lesion was detected at more than one time point, the earliest time point was used.
Time Frame: At 0.5, 1, 2, and 4 hour post-injection on Day 0
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ITT Population (Day 0)
Number analyzed (Participants) | 12
Participants
  Total: At 0.5 hour | 5
  Total: At 1 hour | 3
  Total: At 2 hour | 4
  Total: At 4 hour | 0
  Bone: number analyzed (Participants) | 2
  Bone: At 0.5 hour | 2
  Bone: At 1 hour | 0
  Bone: At 2 hour | 0
  Bone: At 4 hour | 0
  Liver: number analyzed (Participants) | 9
  Liver: At 0.5 hour | 2
  Liver: At 1 hour | 3
  Liver: At 2 hour | 4
  Liver: At 4 hour | 0
  Lung: number analyzed (Participants) | 0
  Lymph node: number analyzed (Participants) | 7
  Lymph node: At 0.5 hour | 7
  Lymph node: At 1 hour | 0
  Lymph node: At 2 hour | 0
  Lymph node: At 4 hour | 0
  Mamma: number analyzed (Participants) | 0
  Pancreas: number analyzed (Participants) | 1
  Pancreas: At 0.5 hour | 1
  Pancreas: At 1 hour | 0
  Pancreas: At 2 hour | 0
  Pancreas: At 4 hour | 0
  Peritoneum: number analyzed (Participants) | 1
  Peritoneum: At 0.5 hour | 1
  Peritoneum: At 1 hour | 0
  Peritoneum: At 2 hour | 0
  Peritoneum: At 4 hour | 0
  Small bowel: number analyzed (Participants) | 3
  Small bowel: At 0.5 hour | 3
  Small bowel: At 1 hour | 0
  Small bowel: At 2 hour | 0
  Small bowel: At 4 hour | 0
  Thyroid gland: number analyzed (Participants) | 0

13. Secondary Outcome: Number of Participants at Each Time Point With the Highest Mean 3D-SUV-R Tumor Value
Description: The time point with the highest mean 3D-SUV-R per tissue location were determined. If the highest mean 3D-SUV-R was detected at more than one time point, the earliest time point was used.
Time Frame: At 0.5, 1, 2, and 4 hour post-injection on Day 0
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ITT Population (Day 0)
Number analyzed (Participants) | 11
Participants
  Bone (RT: Bone): number analyzed (Participants) | 2
  Bone (RT: Bone): At 0.5 hour | 1
  Bone (RT: Bone): At 1 hour | 0
  Bone (RT: Bone): At 2 hour | 1
  Bone (RT: Bone): At 4 hour | 0
  Bone (RT: Muscle): number analyzed (Participants) | 2
  Bone (RT: Muscle): At 0.5 hour | 1
  Bone (RT: Muscle): At 1 hour | 0
  Bone (RT: Muscle): At 2 hour | 1
  Bone (RT: Muscle): At 4 hour | 0
  Liver (RT: Liver): number analyzed (Participants) | 9
  Liver (RT: Liver): At 0.5 hour | 0
  Liver (RT: Liver): At 1 hour | 4
  Liver (RT: Liver): At 2 hour | 2
  Liver (RT: Liver): At 4 hour | 3
  Liver (RT: Muscle): number analyzed (Participants) | 9
  Liver (RT: Muscle): At 0.5 hour | 2
  Liver (RT: Muscle): At 1 hour | 5
  Liver (RT: Muscle): At 2 hour | 2
  Liver (RT: Muscle): At 4 hour | 0
  Lymph node (RT: Lymph node): number analyzed (Participants) | 7
  Lymph node (RT: Lymph node): At 0.5 hour | 2
  Lymph node (RT: Lymph node): At 1 hour | 1
  Lymph node (RT: Lymph node): At 2 hour | 2
  Lymph node (RT: Lymph node): At 4 hour | 2
  Lymph node (RT: Muscle): number analyzed (Participants) | 7
  Lymph node (RT: Muscle): At 0.5 hour | 1
  Lymph node (RT: Muscle): At 1 hour | 5
  Lymph node (RT: Muscle): At 2 hour | 1
  Lymph node (RT: Muscle): At 4 hour | 0
  Mamma (RT: Mamma): number analyzed (Participants) | 0
  Mamma (RT: Muscle): number analyzed (Participants) | 0
  Peritoneum (RT: Peritoneum): number analyzed (Participants) | 1
  Peritoneum (RT: Peritoneum): At 0.5 hour | 0
  Peritoneum (RT: Peritoneum): At 1 hour | 0
  Peritoneum (RT: Peritoneum): At 2 hour | 1
  Peritoneum (RT: Peritoneum): At 4 hour | 0
  Peritoneum (RT: Muscle): number analyzed (Participants) | 1
  Peritoneum (RT: Muscle): At 0.5 hour | 0
  Peritoneum (RT: Muscle): At 1 hour | 1
  Peritoneum (RT: Muscle): At 2 hour | 0
  Peritoneum (RT: Muscle): At 4 hour | 0
  Small bowel (RT: Small bowel): number analyzed (Participants) | 3
  Small bowel (RT: Small bowel): At 0.5 hour | 1
  Small bowel (RT: Small bowel): At 1 hour | 2
  Small bowel (RT: Small bowel): At 2 hour | 0
  Small bowel (RT: Small bowel): At 4 hour | 0
  Small bowel (RT: Muscle): number analyzed (Participants) | 3
  Small bowel (RT: Muscle): At 0.5 hour | 0
  Small bowel (RT: Muscle): At 1 hour | 3
  Small bowel (RT: Muscle): At 2 hour | 0
  Small bowel (RT: Muscle): At 4 hour | 0

14. Secondary Outcome: Best Diagnostic Scan Assessment
Description: The assessment of every diagnostic 68Ga-OPS202 PET/CT scan of session 2 was rated by the reader from 1 to 5, where 1=worst diagnostic scan and 5=best diagnostic scan. Higher score indicates a better scan.
Time Frame: At 0.5, 1, 2, and 4 hour post-injection on Day 0 and 1 hour post-injection on Day 21
Population: as for outcome 4
Measure: Median (Full Range); unit: score on a scale
Arm/Group | ITT Population (Day 0) | ITT Population (Day 21)
Number analyzed (Participants) | 12 | 12
score on a scale
  At 0.5 hour: number analyzed (Participants) | 12 | 0
  At 0.5 hour | 4.0 [2 to 5] |
  At 1 hour | 5.0 [3 to 5] | 5.0 [3 to 5]
  At 2 hour: number analyzed (Participants) | 12 | 0
  At 2 hour | 4.5 [3 to 5] |
  At 4 hour: number analyzed (Participants) | 12 | 0
  At 4 hour | 2.0 [1 to 4] |

ADVERSE EVENTS:
Time Frame: From start of IP administration to end of the study visit (approximately 28 to 36 days).
Description: The SAF included all participants of the FAS who received the IP, regardless of any protocol deviations.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 6/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=12)
Urinary tract infection (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes